CLINICAL TRIAL: NCT07152834
Title: Evaluation of the Relationship Between Dyspnoea and Functional Airway Obstruction in Alpha-1 Antitrypsin Deficiency: A Prospective, Case-Control, Analytical Study
Brief Title: Screening for Alpha-1 Antitrypsin Deficiency in Patients With Airway Obstruction
Acronym: AATD-SAO
Status: Recruiting | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: PROGENIKA BIOPHARMA, A GRIFOLS Company (Unknown)
Responsible Party: Principal Investigator, Ozlem Sengoren Dikis, Associate Professor, Muğla Sıtkı Koçman University
Other Study IDs: Alpha1
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Alpha 1-antitrypsin Deficiency (AATD)
Keywords: Alpha 1-Antitrypsin Deficiency; Airway Obstruction; PRISm
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Airway Obstruction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The following biological samples will be retained for the duration of the study:
  Residual serum from routine clinical blood samples, aliquoted and stored in polypropylene cryotubes at -80°C for Alpha-1 Antitrypsin (AAT) level quantification.
  Capillary whole blood collected via finger prick, stored on filter paper or in micro-containers, for DNA extraction and SERPINA1 genotyping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRISm: Patients with a post-bronchodilator FEV1/FVC ratio ≥ 0.70, FEV1 < 80
  Interventions: Diagnostic Test: Blood Sampling
- Normal PFT: Patients with a post-bronchodilator FEV1/FVC ratio ≥ 0.70, FEV1 ≥ 80
  Interventions: Diagnostic Test: Blood Sampling

INTERVENTIONS:
Diagnostic Test: Blood Sampling — For AAT Level: Residual serum from routine blood samples drawn for standard clinical care will be aliquoted into polypropylene cryotubes.
  For Genetic Testing: A separate capillary blood sample will be obtained via finger prick using a sterile lancet and collected on a designated filter paper.

SUMMARY:
Brief Summary:

This study aims to find out if a genetic condition called Alpha-1 Antitrypsin Deficiency (AATD) is more common in people who have shortness of breath and signs of airway obstruction on their breathing tests.

Alpha-1 antitrypsin (AAT) is a protein that protects the lungs from damage. AATD is an inherited condition where the body does not make enough of this protein, which can lead to lung diseases like emphysema, especially in smokers.

Investigators hypothesize that low AAT levels or related genetic mutations may be a contributing factor to airway obstruction in patients complaining of shortness of breath.

To test this, investigators will recruit patients from our outpatient clinic who are being evaluated for shortness of breath and are having a standard breathing test (spirometry). Investigators will measure their AAT levels and test for the most common genetic mutations that cause AATD using a small blood sample. Investigators will then compare the AAT levels and genetic results between different groups of patients, such as smokers and non-smokers with and without airway obstruction. Investigators will also see if the severity of a patient's shortness of breath is related to their AAT levels.

The goal is to improve the detection of AATD in this patient population, which could lead to better diagnoses and specific treatments for those who have this condition.

DETAILED DESCRIPTION:
1. Study Objectives and Rationale Alpha-1 Antitrypsin Deficiency (AATD) is a significantly underdiagnosed hereditary disorder that predisposes individuals to early-onset emphysema and chronic obstructive pulmonary disease (COPD), particularly in smokers. The primary objective of this single-center, cross-sectional, analytical study is to determine the prevalence of both quantitative (serum level) and qualitative (genetic mutation) AATD in a targeted, high-risk population: patients presenting to a pulmonary outpatient clinic with shortness of breath (dyspnea) and found to have functional airway obstruction on spirometry.

   The study operates on the hypothesis that a subset of patients with airway obstruction, especially those with an early onset or a disproportionate severity of disease relative to their smoking history, may have undiagnosed AATD. By systematically screening this population using both serum level analysis and genetic testing, we aim to identify a previously undetected patient cohort, enabling earlier intervention, family screening, and specific management strategies.
2. Study Design and Methodology This is a prospective, case-control, analytical study conducted at the Chest Diseases Outpatient Clinic of Muğla Training and Research Hospital.

Participant Flow:

1. Screening & Identification: Consecutive patients presenting with a chief complaint of dyspnea who are scheduled for routine diagnostic spirometry as part of standard clinical care will be assessed for eligibility.
2. Informed Consent: Eligible patients will be provided with a detailed informed consent form explaining the study's purpose, procedures, risks, and benefits.
3. Group Allocation: Following spirometry, participants will be allocated into two groups based on their test results:

   Case Group (PRISm): Patients with a post-bronchodilator FEV1/FVC ratio ≥ 0.70, FEV1 < 80 Control Group (No Airway Obstruction): Patients with a post-bronchodilator FEV1/FVC ratio ≥ 0.70, FEV1 ≥ 80
4. Data and Sample Collection: All participants will undergo:

   Clinical Assessment: Recording of mMRC dyspnea scale and detailed smoking history.

   Blood Sampling:

   For AAT Level: Residual serum from routine blood samples drawn for standard clinical care will be aliquoted into polypropylene cryotubes.

   For Genetic Testing: A separate capillary blood sample will be obtained via finger prick using a sterile lancet and collected on a designated filter paper.
5. Blinding: Laboratory personnel performing the AAT level assays and genetic analyses will be blinded to the participant's group assignment (case or control) and clinical data.

Laboratory Methods:

AAT Serum Level Measurement: Serum AAT concentrations will be quantified using a validated immunoturbidimetric assay on an automated clinical chemistry analyzer.

Genetic Analysis: DNA will be extracted from the capillary blood samples. Genotyping for the most common pathogenic *SERPINA1* alleles (e.g., PI*S, PI*Z) will be performed using a real-time polymerase chain reaction (RT-PCR) based method.

3. Data Management and Quality Assurance

Data Collection and Source Documents: Clinical data (spirometry results, mMRC, smoking history) will be recorded directly into a structured electronic Case Report Form (eCRF). Spirometry equipment will be calibrated daily according to American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines. Source documents include hospital medical records and laboratory information system reports.

4. Statistical Analysis Plan A review of the national and international literature revealed no prior studies specifically investigating the clinical characteristics of airway obstruction in relation to alpha-1 antitrypsin genetic mutations and/or levels, underscoring the novelty of this research.

The sample size calculation was performed using the G*Power 3.1.2 software. Based on FEV1 measurements (mean ± SD = 56 ± 13) reported in a reference study of dyspnoeic patients, the effect size was calculated as 0.1538462. This calculation determined that a minimum of 334 participants per group would be required to achieve 80% statistical power with a 5% margin of error (alpha = 0.05). Anticipating a potential 10% dropout rate, the target sample size was increased to at least 367 patients for the case group and 367 matched controls for the control group.

All statistical analyses will be conducted using IBM SPSS Statistics for Windows, Version 27.0 (Armonk, NY: IBM Corp.). The normality of distribution for quantitative variables will be assessed using the Kolmogorov-Smirnov test. For comparisons between independent groups:

Normally distributed variables will be analyzed using the Independent Samples t-test (for two groups) or One-Way ANOVA (for more than two groups).

Non-normally distributed variables will be analyzed using the Mann-Whitney U test (for two groups) or the Kruskal-Wallis H test (for more than two groups).

The relationship between qualitative variables will be investigated using Chi-square analysis. Correlations between quantitative variables will be examined using Pearson's correlation coefficient for normally distributed data or Spearman's rank correlation coefficient for non-normal data.

To identify factors independently associated with the presence of breathlessness (dyspnea), multivariate analyses will be employed. This will include data-structure-appropriate binary logistic regression models. Additionally, advanced analytical techniques such as decision tree methods (e.g., C&RT, C4.5) may be applied for predictive modeling and pattern recognition.

Descriptive statistics will be reported as follows:

Normally distributed quantitative variables: Mean ± Standard Deviation. Non-normally distributed quantitative variables: Median (25th - 75th percentile) or Median (Minimum - Maximum).

Categorical variables: Frequency (n, %). A p-value of less than 0.05 will be considered statistically significant for all analyses.

**5. Ethical and Operational Considerations** The study protocol has been approved by the Muğla Sıtkı Koçman University Local Ethics Committee. All biological samples will be stored anonymized and coded in a dedicated -80°C freezer with restricted access. Samples will be destroyed according to ethical guidelines upon study completion.

ELIGIBILITY:
Inclusion Criteria:

* Achieve a post-bronchodilator FEV1/FVC ratio of 70 or above in the respiratory function test.
* Be able to speak and understand Turkish.
* Have the mental and cognitive capacity to understand the questions asked.

Exclusion Criteria:

* Renal dysfunction; acute inflammation; rheumatological, haematological, or liver diseases; COPD; asthma; bronchiectasis; and a history of malignancy.
* Pregnant women and users of oral contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of consecutive adult patients presenting with a primary complaint of dyspnoea (shortness of breath) at the Chest Diseases Outpatient Clinic of Muğla Training and Research Hospital in Turkey. These patients will be referred for routine diagnostic pulmonary function testing (spirometry) as part of their standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 734 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Alpha-1 Antitrypsin Deficiency (AATD) | Day 1
  The prevalence of Alpha-1 Antitrypsin Deficiency (AATD) is defined as the proportion of participants in each group who test positive for the condition. AATD is diagnosed by either:
  Genetic Analysis: Identification of a pathogenic SERPINA1 mutation (e.g., PIZ or PIS allele) via PCR-based genotyping of a capillary blood sample.
  Serum Level Analysis: A serum AAT concentration below 0.9 g/L, measured using an immunoturbidimetric assay on a residual serum sample from routine blood work.
  The difference in prevalence rates between the case and control groups will be statistically compared.

SECONDARY OUTCOMES:
Correlation between AATD and smoking status. | Day 1
  The correlation between AATD and smoking habits will be analyzed by comparing the % of patients with AATD (as defined above) across different smoking status categories (never-smoker, former smoker, current smoker) within the study groups. Smoking history is quantified by patient-reported pack-years.

OTHER OUTCOMES:
Correlation between dyspnea severity and AAT level. | Day 1
  The correlation between dyspnea severity and AAT level will be assessed by calculating the correlation coefficient between the quantitative serum AAT level (g/L) and the mMRC (Modified Medical Research Council) dyspnea scale score. The mMRC is a 5-point scale (0-4) where 0 means breathlessness only with strenuous exercise and 4 means too breathless to leave the house or breathless when dressing. A higher score indicates worse dyspnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) that underlie the results reported in publications from this study will not be made publicly available. This decision is based on several factors: the data contain sensitive genetic and health information, the informed consent process obtained from participants did not include provisions for public data sharing, and the current ethical approval and local data protection regulations at Muğla Training and Research Hospital restrict the public sharing of such identifiable personal health data. Requests for anonymized data may be considered on a case-by-case basis for legitimate research purposes, subject to a formal data sharing agreement and approval from the local ethics committee.